CLINICAL TRIAL: NCT00213200
Title: Systemic Analgesia and Local Anaesthesia for Percutaneous Venous Catheter Placement in Preterm Neonates
Brief Title: Intravenous and Topical Analgesics for Procedural Pain in Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Society of Hospital Pharmacists (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0019990251
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2005-09

CONDITIONS: Pain; Infant, Newborn
Keywords: pain; analgesia; morphine; amethocaine; neonate
MeSH Terms: conditions — Pain; Agnosia | interventions — Morphine; Tetracaine

INTERVENTIONS:
Drug: morphine, amethocaine

SUMMARY:
This study will test which type of pain medication is best for the management of pain in newborn preterm and full-term infants having a deep intravenous cannula inserted. It will compare the effectiveness of intravenous morphine alone, a local anaesthetic cream (amethocaine) alone, and both medications together. It will also determine the safety of both medications.

ELIGIBILITY:
Inclusion Criteria:

* preterm and full-term infants in the NICU requiring a percutaneous central venous catheter
* ventilatory support in the form of conventional ventilation, Continuous Positive Air Pressure (CPAP) or High Frequency Oscillation(HFO)

Exclusion Criteria:

* seizures
* receiving muscle relaxants
* skin disorders causing disruption of stratum corneum

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108
Dates: Start 2003-07; Study Completion 2005-06

PRIMARY OUTCOMES:
- Facial grimacing, as assessed by brow bulge, at the time of the procedure, compared among groups

SECONDARY OUTCOMES:
heart rate at the time of procedure
oxygen saturation at the time of procedure
local skin reactions at the time of procedure
blood pressure for 24 hours post procedure
ventilatory support for 24 hours post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Result] Taddio A, Lee C, Yip A, Parvez B, McNamara PJ, Shah V. Intravenous morphine and topical tetracaine for treatment of pain in [corrected] neonates undergoing central line placement. JAMA. 2006 Feb 15;295(7):793-800. doi: 10.1001/jama.295.7.793. PMID 16478902